CLINICAL TRIAL: NCT00152230
Title: A Randomized Controlled Study of Postoperative Adjuvant Chemotherapy of UFT Compared With Surgery Alone in Patients With Dukes C Colorectal Cancer (NSAS-CC)
Brief Title: A Randomized Controlled Study of Postoperative Adjuvant Chemotherapy of Uracil- Tegafur (UFT) Compared With Surgery Alone (NSAS-CC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Taiho Pharmaceutical Co., Ltd., Taiho Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01023002
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Tegafur; Uracil; Surgical Procedures, Operative

ARMS (2):
- 1 (Experimental): UFT (uracil, tegafur)
  Interventions: Drug: UFT (uracil, tegafur)
- 2 (Other): Surgery alone
  Interventions: Procedure: Surgery alone

INTERVENTIONS:
Drug: UFT (uracil, tegafur) — to receive oral uracil-tegafur 400 mg square meter for one year
  Arms: 1
Procedure: Surgery alone — Standardized mesorectal excision with selective lateral pelvic lymphadenectomy of stage III rectal cancer.
  Arms: 2

SUMMARY:
This is a controlled study designed to compare relapse-free survival and overall survival in patients receiving UFT with those in patients receiving surgery alone. Patients will be randomly assigned to surgery alone or surgery followed by UFT within 6 weeks after curative resection. To assess treatment efficacy, data on recurrence and survival will be collected for 5 years after enrollment of the last patient. To evaluate safety, data on adverse events will be collected for 12 months after the start of treatment.Evaluations will be separately done for colon cancer and rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 75
* Performance status 0 , 1, or 2 (ECOG)
* Hematopoietic WBC ≥ 4,000/mm^3 Platelet ≥ 100,000/mm^3
* Hepatic AST and ALT ≤ 2 times upper limit of normal(ULN) Total bilirubin ≤ 1.2mg/dL
* Renal BUN ≤ 25mg/dL Creatinine ≤ 1.5mg/dL

Exclusion Criteria:

* Prior anticancer treatment

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 1996-10; Primary Completion 2006-03 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival and overall survival | every course for first three courses, then every other course

SECONDARY OUTCOMES:
Adverse events | any time

CONTACTS AND LOCATIONS:
Overall Officials: Shigeaki Yoshida, MD, Principal Investigator — National Cancer Center Hospital East
Locations (1):
- National Cancer Center Hospital East, 6-5-1, Kashiwanoha, Kashiwa, Chiba, Japan

REFERENCES:
- [Background] Hamaguchi T, Shirao K, Moriya Y, Yoshida S, Kodaira S, Ohashi Y; NSAS-CC Group. Final results of randomized trials by the National Surgical Adjuvant Study of Colorectal Cancer (NSAS-CC). Cancer Chemother Pharmacol. 2011 Mar;67(3):587-96. doi: 10.1007/s00280-010-1358-1. Epub 2010 May 19. PMID 20490797
- [Result] Akasu T, Moriya Y, Ohashi Y, Yoshida S, Shirao K, Kodaira S; National Surgical Adjuvant Study of Colorectal Cancer. Adjuvant chemotherapy with uracil-tegafur for pathological stage III rectal cancer after mesorectal excision with selective lateral pelvic lymphadenectomy: a multicenter randomized controlled trial. Jpn J Clin Oncol. 2006 Apr;36(4):237-44. doi: 10.1093/jjco/hyl014. Epub 2006 May 4. PMID 16675478